CLINICAL TRIAL: NCT06146868
Title: Gerontechnology Evaluation Framework: Outcome Validation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: Gerontechnology Platform, The Social Innovation and Entrepreneurship Development Fund (Unknown)
Responsible Party: Principal Investigator, Dr. Derek Yee-Tak Cheung, Assistant Professor, The University of Hong Kong
Other Study IDs: Gerontechnology Outcome
Record Dates: First submitted 2023-11-17; First posted 2023-11-27 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Technology
Keywords: Gerontechnology; Outcome indicators

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Staff: A cross-sectional survey will be conducted.
  Interventions: Other: Doing questionnaire
- User: A cross-sectional survey will be conducted.
  Interventions: Other: Doing questionnaire
- Caregiver: A cross-sectional survey will be conducted.
  Interventions: Other: Doing questionnaire
- Supplier: A cross-sectional survey will be conducted.
  Interventions: Other: Doing questionnaire

INTERVENTIONS:
Other: Doing questionnaire — Participants will provide their opinions in a questionnaire

SUMMARY:
The project aims to validate the evaluation indicators applicability of 9 Gerontechnology Evaluation Frameworks. The outcome is the perceived importance of the evaluation indicators described in the 9 Evaluation Frameworks. Participants will be invited to complete a questionnaire indicating the importance of the outcomes.

DETAILED DESCRIPTION:
This study is a cross-sectional survey. 165 to 300 participants will be recruited to complete a questionnaire. For each product theme that they are familiar with, they will rate anonymously the perceived importance of the evaluation indicators on a 5-point Likert scale, give reasons for their ratings and suggest revisions.

Participants will be recruited through convenience sampling in 3 subgroups, including (1) members of Gerontechnology Application and Testing Working Group under Gerontechnology Platform, (2) successful applicants of Innovation and Technology Fund for buying gerontechnology products under the 9 themes, and (3) visitors of Gerontech and Innovation Expo. It is expected that 35% participants will be recruited in subgroup 1, 5% in subgroup 2, and 60% in subgroup 3.

Gerontechnology Platform will invite (1) its members of Gerontechnology Application and Testing Working Group, who are the Users, Caregivers, Staff and Suppliers of gerontechnology products, to fill in the questionnaire online. 3 email reminders will be sent to remind them to complete the questionnaire. (2) The list of successful applicants of Innovation and Technology Fund who applied for the product themes covered in the 9 Evaluation Frameworks will be downloaded from the Social Welfare Department website and their Staff will be invited to fill in the questionnaire online. (3) In Gerontech and Innovation Expo, which is a local exhibition that provides a platform for stakeholders to discuss and collaborate for broader adoption of gerontechnology, research staff will approach all visitors of the Gerontechnology Platform booth. The visitors who fulfil the inclusion and exclusion criteria will be invited to complete the questionnaire.

To ensure the validity of their responses, they will only answer the questionnaire items of the themes they have known, have used, or are most interested. For each product theme that they are familiar with, they will rate anonymously the perceived importance of the evaluation indicators on a 5-point Likert scale, give reasons for their ratings and suggest revisions. Their voluntary written consent will be sought before they complete the questionnaire. Each questionnaire will take around 5 - 10 minutes.

ELIGIBILITY:
Inclusion Criteria:

* People in one of these categories: Working or has worked in a social service setting for the elderly or person with disability (Staff), an elderly aged 60 or above (User), a person with physical or disability (User), an informal caregiver for an elderly or a person with disability (Caregiver), or belonging to a company/or that has developed or retailed gerontechnology products (Supplier)

Exclusion Criteria:

* Unable to read or write in Chinese

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Stakeholders of gerontechnology in Hong Kong
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Degree of importance on indicators of fall prevention Framework | 3 months
  The level of agreement on indicators of fall prevention Framework. The opinions will be categorized into four levels of consensus according to the central tendency, level of dispersion, and the rated level of importance (Shi et al., 2022). The consensus levels are defined as: very high consensus (median = 5, inter-quartile range (IQR) = 0, rating score of 4/5 ≥ 80%); high consensus (median = 5, IQR = 1, rating score of 4/5 ≥ 80%); moderate consensus (median = 4-5, IQR = 1, rating score 4/5 ≥ 75%), and low consensus (median ≤ 4, IQR ≤ 2, rating score 4/5 < 75%).
Degree of importance on indicators of health monitoring Framework | 3 months
  The level of agreement on indicators of health monitoring Framework. The opinions will be categorized into four levels of consensus according to the central tendency, level of dispersion, and the rated level of importance (Shi et al., 2022). The consensus levels are defined as: very high consensus (median = 5, inter-quartile range (IQR) = 0, rating score of 4/5 ≥ 80%); high consensus (median = 5, IQR = 1, rating score of 4/5 ≥ 80%); moderate consensus (median = 4-5, IQR = 1, rating score 4/5 ≥ 75%), and low consensus (median ≤ 4, IQR ≤ 2, rating score 4/5 < 75%).
Degree of importance on indicators of transfer and lifting Framework | 3 months
  The level of agreement on indicators of transfer and lifting Framework. The opinions will be categorized into four levels of consensus according to the central tendency, level of dispersion, and the rated level of importance (Shi et al., 2022). The consensus levels are defined as: very high consensus (median = 5, inter-quartile range (IQR) = 0, rating score of 4/5 ≥ 80%); high consensus (median = 5, IQR = 1, rating score of 4/5 ≥ 80%); moderate consensus (median = 4-5, IQR = 1, rating score 4/5 ≥ 75%), and low consensus (median ≤ 4, IQR ≤ 2, rating score 4/5 < 75%).
Degree of importance on indicators of hygiene management Framework | 3 months
  The level of agreement on indicators of hygiene management Framework. The opinions will be categorized into four levels of consensus according to the central tendency, level of dispersion, and the rated level of importance (Shi et al., 2022). The consensus levels are defined as: very high consensus (median = 5, inter-quartile range (IQR) = 0, rating score of 4/5 ≥ 80%); high consensus (median = 5, IQR = 1, rating score of 4/5 ≥ 80%); moderate consensus (median = 4-5, IQR = 1, rating score 4/5 ≥ 75%), and low consensus (median ≤ 4, IQR ≤ 2, rating score 4/5 < 75%).
Degree of importance on indicators of communication Framework | 3 months
  The level of agreement on indicators of communication Framework. The opinions will be categorized into four levels of consensus according to the central tendency, level of dispersion, and the rated level of importance (Shi et al., 2022). The consensus levels are defined as: very high consensus (median = 5, inter-quartile range (IQR) = 0, rating score of 4/5 ≥ 80%); high consensus (median = 5, IQR = 1, rating score of 4/5 ≥ 80%); moderate consensus (median = 4-5, IQR = 1, rating score 4/5 ≥ 75%), and low consensus (median ≤ 4, IQR ≤ 2, rating score 4/5 < 75%).
Degree of importance on indicators of anti-wandering Framework | 3 months
  The level of agreement on indicators of anti-wandering Framework. The opinions will be categorized into four levels of consensus according to the central tendency, level of dispersion, and the rated level of importance (Shi et al., 2022). The consensus levels are defined as: very high consensus (median = 5, inter-quartile range (IQR) = 0, rating score of 4/5 ≥ 80%); high consensus (median = 5, IQR = 1, rating score of 4/5 ≥ 80%); moderate consensus (median = 4-5, IQR = 1, rating score 4/5 ≥ 75%), and low consensus (median ≤ 4, IQR ≤ 2, rating score 4/5 < 75%).
Degree of importance on indicators of air quality sensor Framework | 3 months
  The level of agreement on indicators of air quality sensor Framework. The opinions will be categorized into four levels of consensus according to the central tendency, level of dispersion, and the rated level of importance (Shi et al., 2022). The consensus levels are defined as: very high consensus (median = 5, inter-quartile range (IQR) = 0, rating score of 4/5 ≥ 80%); high consensus (median = 5, IQR = 1, rating score of 4/5 ≥ 80%); moderate consensus (median = 4-5, IQR = 1, rating score 4/5 ≥ 75%), and low consensus (median ≤ 4, IQR ≤ 2, rating score 4/5 < 75%).
Degree of importance on indicators of feeding tools Framework | 3 months
  The level of agreement on indicators of feeding tools Framework. The opinions will be categorized into four levels of consensus according to the central tendency, level of dispersion, and the rated level of importance (Shi et al., 2022). The consensus levels are defined as: very high consensus (median = 5, inter-quartile range (IQR) = 0, rating score of 4/5 ≥ 80%); high consensus (median = 5, IQR = 1, rating score of 4/5 ≥ 80%); moderate consensus (median = 4-5, IQR = 1, rating score 4/5 ≥ 75%), and low consensus (median ≤ 4, IQR ≤ 2, rating score 4/5 < 75%).
Degree of importance on indicators of cognitive training and stimulation Framework | 3 months
  The level of agreement on indicators of cognitive training and stimulation Framework. The opinions will be categorized into four levels of consensus according to the central tendency, level of dispersion, and the rated level of importance (Shi et al., 2022). The consensus levels are defined as: very high consensus (median = 5, inter-quartile range (IQR) = 0, rating score of 4/5 ≥ 80%); high consensus (median = 5, IQR = 1, rating score of 4/5 ≥ 80%); moderate consensus (median = 4-5, IQR = 1, rating score 4/5 ≥ 75%), and low consensus (median ≤ 4, IQR ≤ 2, rating score 4/5 < 75%).

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be available

REFERENCES:
- [Background] Shi C, Wong GHY, Choy JCP, Wong KKY, Lum TYS, Yu DSF. Are we on the same page? Multiple stakeholders and service users priorities for dementia care and policy: A Delphi study. Int J Nurs Stud. 2022 Sep;133:104300. doi: 10.1016/j.ijnurstu.2022.104300. Epub 2022 May 28. PMID 35751948